CLINICAL TRIAL: NCT04983615
Title: Opioid vs. Benzodiazepine-based Sedation for Mechanically Ventilated Patients in the Internal Medicine Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0114-21-MMC
Record Dates: First submitted 2021-07-25; First posted 2021-07-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Mechanically Ventilated Patients
Keywords: opioid-based sedation, delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl-based sedation group (Experimental)
  Interventions: Drug: fentanyl-based sedation
- midazolam-based sedation group (Active Comparator)
  Interventions: Drug: midazolam-based sedation

INTERVENTIONS:
Drug: fentanyl-based sedation — fentanyl-based sedation instead of midazolam-based sedation in ventilated patients
  Arms: fentanyl-based sedation group
Drug: midazolam-based sedation — midazolam-based sedation
  Arms: midazolam-based sedation group

SUMMARY:
Opioid-based sedation as a first line in mechanically ventilated patients has been considered the "gold standard" in intensive care unit patients around the world for several decades. Advantages of opiate-based sedation, compared to benzodiazepine-based sedation, which has been used in the past, include a reduction in delirium scores, better pain control, decreasing the time between cessation of sedation and patient awakening, and decreasing the time between cessation of sedation and extubation, with decreased ICU admission times.

In most Western European countries, as well as in the United States, there are almost no mechanically ventilated patients hospitalized outside the intensive care unit. In a few countries, including Japan and Israel, mechanically ventilated patients are also hospitalized outside of intensive care units, as part of internal or surgical wards. Contrary to the vast knowledge accumulated regarding different sedation methods in ventilated patients in intensive care units, there are almost no studies that have evaluated different sedation methods in ventilated patients hospitalized in non-intensive care wards. Thus, while there is consensus on the benefits of opioid-based sedation in intensive care units, there is insufficient information to recommend the preferred sedation method in non-ICU wards.

For various reasons, in a large number of the internal medicine wards of hospitals in Israel, the common sedation practice for ventilated patients is still benzodiazepine-based sedation. In the past year, a pilot program was initiated in Internal Medicine Department A at Meir Hospital in Kfar Saba, in which a new protocol for opioid-based sedation in ventilated patients was implemented.

The protocol is based on the continuous intravenous infusion of fentanyl as the first line of treatment for sedation in ventilated patients only. If the sedation-agitation level (as measured by the RASS score) did not match the target RASS score set by the attending physician, a dose up to a maximum limit could be increased according to the protocol. Second-line sedation drugs were addition of continuous intravenous infusion of midazolam (in addition to fentanyl) in hemodynamically stable patients, or addition of continuous intravenous infusion of ketamine in unstable patients. In stable patients who did not reach the desired RASS level under continuous infusion of fentanyl and midazolam, ketamine could be added as a third line drug, in addition to fentanyl and midazolam.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18-99 who were admitted to Internal Medicine Department A at Meir Hospital in Kfar Saba from January 2020 to January 2021 (inclusive), and required mechanical ventilation.

-

Exclusion Criteria: Patients who were sedated and ventilated for palliative care only without any fututre plan for weaning them of ventilation, or patients in whom there was a deviation from the treatment protocol

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
RASS score | 1 year
  comparison of delirium score between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Sara Dichtwald, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No